CLINICAL TRIAL: NCT02174770
Title: Blood Flow Restriction Training Versus Standard Physical Therapy in Post-Operative and Post-Traumatic Rehabilitation Patients
Brief Title: Blood Flow Restriction Training in Rehabilitation Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of resources
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Christina Hylden, Orthopaedic Surgery Resident, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 395166; 397709 (Other Grant/Funding Number: AAMTI)
Record Dates: First submitted 2014-06-23; First posted 2014-06-26 (Estimated); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Anterior Cruciate Ligament Reconstruction; Volumetric Muscle Loss; Chronic Thigh Muscle Weakness; Knee Arthroscopy
MeSH Terms: interventions — Blood Flow Restriction Therapy; Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- ACL BFR group (Experimental): This group is patients with post-op from ACL reconstruction who are randomized into the blood flow restriction arm. They will receive BFR strength training as part of their post-operative physical therapy program for two months during normal post-op rehab.
  Interventions: Other: Blood Flow Restriction (BFR) Training
- ACL Standard Therapy (Active Comparator): This group is patients with post-op from ACL reconstruction who are randomized into the standard therapy arm. They will receive ACSM guided-strength training as part of their post-operative physical therapy program.
  Interventions: Other: Standard ACSM-guided strength training
- Chronic Muscle Weakness (Other): This is a crossover group where all subjects will be randomized to begin with either standard or blood flow restriction therapy for 4 weeks. After completion of the initial training, each subject will be switched to the opposite in an AB/BA crossover design.
  Interventions: Other: Blood Flow Restriction (BFR) Training; Other: Standard ACSM-guided strength training
- Knee Arthroscopy BFR (Experimental): This group is patients with post-op from soft-tissue only knee arthroscopy who are randomized into the blood flow restriction arm. They will receive BFR strength training as part of their post-operative physical therapy program for two months during normal post-op rehab.
  Interventions: Other: Blood Flow Restriction (BFR) Training
- Knee Arthroscopy Standard (Active Comparator): This group is patients with post-op from soft-tissue only knee arthroscopy who are randomized into the standard physical therapy arm. They will receive ACSM-guided strength training as part of their post-operative physical therapy program during normal post-op rehab.
  Interventions: Other: Standard ACSM-guided strength training

INTERVENTIONS:
Other: Blood Flow Restriction (BFR) Training — This is a modality of physical therapy where during low-load resistance activity, the venous return of blood from an extremity is limited only during the duration of the exercise. This can be accomplished through multiple means. For the purposes of our study, we will use an inflatable tourniquet.
  Other Names: Low resistance training; Occlusion training
  Arms: ACL BFR group; Chronic Muscle Weakness; Knee Arthroscopy BFR
Other: Standard ACSM-guided strength training — This is the standard protocol to be used for post-operative and other physical therapy patients for rehabilitation. It includes the use of American College of Sports Medicine-guidelines for how much weight to use during the strength training portion of the rehabilitation.
  Other Names: physical therapy
  Arms: ACL Standard Therapy; Chronic Muscle Weakness; Knee Arthroscopy Standard

SUMMARY:
Occlusion training, resistance exercise performed with a specialized venous tourniquet, leads to beneficial changes in muscle at low resistance and minimal stress on the nearby joint. This novel resistance training has the potential to greatly improve extremity muscle strength gains for rehabilitation patients who are unable for medical reasons to perform high resistance exercise. Our study will explore this with specific rehabilitation populations: post-operative knee scopes, post-operative anterior cruciate ligament (ACL) reconstruction patients who have acute post-operative changes in thigh muscle function and chronic thigh weakness. The primary outcome is to achieve accelerated functional thigh recovery with outcome measures including thigh strength, validated questionnaires, and validated functional testing. Occlusion training can enhance rehab patients outcomes, reduce the cost of care, and improve the skills and efficiency of care providers.

DETAILED DESCRIPTION:
Occlusion training is the restriction of venous outflow from an extremity with the use of a tourniquet during weight-training or resistance exercises. The technique is a safe and effective method of improving strength through muscle hypertrophy in healthy, active individuals (1-7). The technique has also been shown to be safe and effective in patient populations with various comorbidities (8).These strength gains can be achieved while training with loads as low as 20% of an individual's one repetition maximum (1RM). This is contrary to the American College of Sports Medicine (ACSM) weight-training guidelines that state muscle hypertrophy can only be achieved when an individual lifts loads close to 80% of the 1RM (9).

The purpose of this project is to compare occlusion resistance training to traditional resistance training methods for rehabilitation patients. This will include both an acute post-operative ACL reconstruction cohort and a chronic thigh weakness cohort. Post-operative lower extremity weakness as well as chronic muscle weakness after trauma correlate with lower functional performance.(10,11) We will treat the patients and follow these two cohorts simultaneously.

Specific Aim 1: To determine if occlusion training will accelerate the recovery of thigh muscle function and strength in post-operative anterior cruciate ligament (ACL) reconstruction as compared to a standard post-operative rehabilitation protocol.

Specific Aim 2: To determine if occlusion training will increase quadricep and hamstring muscle function for battlefield wounded warriors with severe thigh weakness as a result of trauma or volumetric muscle loss as compared to standard ACSM resistance training guidelines.

Specific Aim 3: To determine if occlusion training will accelerate the recovery of thigh muscle function and strength in post-operative soft tissue knee arthroscopy as compared to a standard post-operative rehabilitation protocol.

ELIGIBILITY:
Inclusion Criteria:

* One of the following: (1) s/p ACL reconstruction within the last three months prior to initiation of study training, (2) s/p knee arthroscopy within the last 2 weeks prior to initiation of study training, (3) S/p lower extremity trauma, unilateral with thigh weakness of at lest a 20% deficit compared to contralateral side and at least 6 months out from most recent trauma or surgery
* Fluent in English and able to consent

Exclusion Criteria:

* Contralateral lower extremity involvement resulting in less than normal range of motion, muscle strength, or daily pain greater than 5/10.
* Pregnancy, verbal reporting
* Recent history of deep vein thrombosis, within the 12 months or on active treatment
* History of endothelial dysfunction, peripheral vascular disease, hypertension, diabetes, or people prone to capillary ruptures (bruising) (determined by verbal reporting by the patient)
* Active Infection
* Cancer (current diagnosis)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Thigh Muscle Strength | 6 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Center for the Intrepid, Fort Sam Houston, Texas